CLINICAL TRIAL: NCT03147534
Title: Comparison of the InstaTemp MD® Infrared Thermometer With Standard Thermometry in Canadian Routine Clinical Practice
Brief Title: Comparison of Thermometry in Canada for Pediatrics
Acronym: CIT-CRCP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit patients
Sponsor: ARC Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIT-CRCP-001
Record Dates: First submitted 2017-04-19; First posted 2017-05-10 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Healthy; Febrile Illness
MeSH Terms: interventions — Administration, Rectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Children Age 1 month to 2 years (Active Comparator): Collecting temperatures on patients using the ARC InstaTemp MD and a "Welch Allyn" rectal thermometer.
  Interventions: Device: InstaTemp MD; Device: "Welch Allyn", rectal
- Children > 2 to 5 years (Active Comparator): Collecting temperatures on patients using the ARC InstaTemp MD, the "Welch Allyn" rectal and Covidien tympanic thermometer.
  Interventions: Device: InstaTemp MD; Device: "Welch Allyn", rectal; Device: Covidien, tympanic
- Children > 5 to ≤ 10 years (Active Comparator): Collecting temperatures on patients using the ARC InstaTemp MD, the "Welch Allyn" oral and the Covidien tympanic thermometer.
  Interventions: Device: InstaTemp MD; Device: "Welch Allyn", oral; Device: Covidien, tympanic

INTERVENTIONS:
Device: InstaTemp MD — The InstaTemp MD is a hand held electronic infrared thermometer that is intended to accurately measure human body temperature without contact with the human body.
Device: "Welch Allyn", rectal — The "Welch Allyn" rectal thermometer is intended to measure human body temperature.
  Arms: Children > 2 to 5 years; Children Age 1 month to 2 years
Device: "Welch Allyn", oral — The "Welch Allyn" oral thermometer is intended to measure human body temperature.
  Arms: Children > 5 to ≤ 10 years
Device: Covidien, tympanic — The Covidien tympanic thermometer is intended to measure human body temperature.
  Arms: Children > 2 to 5 years; Children > 5 to ≤ 10 years

SUMMARY:
Compare and assess the accuracy and reliability of the InstaTemp MD® device to techniques presently in use for measuring temperature in infants and children in a Canadian clinical setting.

DETAILED DESCRIPTION:
This study is designed as a multi-center study. This study will involve collecting temperatures on patients using the InstaTemp MD® device and the traditional method used in the clinical setting. Reliability and agreement of the InstaTemp MD® will be compared to the current Canadian Paediatric Society's definitely recommended methods of temperature measurement in certain age cohorts of infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Children Age 1 month to ≤ 10 years old
* Male or female
* Subject's parent or legal guardian over the age of 18 years must sign an informed consent form before any study-related procedures are performed
* Subjects who in the opinion of the investigator (or as required by the ethics committee) have the capacity to understand and sign an assent form, must provide written assent

Exclusion Criteria:

* Subjects who in the opinion of the researcher are too agitated, distressed or who are otherwise unable to cooperate with study procedures
* Subjects whose forehead cannot be fully exposed to the ambient condidtions for at least 15 minutes.
* Subjects with signs or recent history of inflammation or infection of the forehead or at the reference clinical test site.
* Subjects currently using cooling blankets or fans
* Subjects with tubes in their ear(s) cannot participate in the tympanic comparison, but this is not exclusionary for InstaTemp MD and definitive comparator (e.g. rectal or oral) measurements.
* Subjects currently receiving treatment with thyroxine, barbiturates, antipsychotics, cortico-steroids (oral iv, or topically applied to forehead)
* Subjects currently alcohol intoxicated
* Subjects with documented illicit durg use in the previous 5 days
* Subjects that have had any hot or cold drinks within 15 minutes prior to a sublingual reading
* Subject is taking any medication that in the opinion of the investigator may alter the temperature of the child
* Subjects participating in a clinical trial of an investigational medicinal product within the last 30 days.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Temperature measurements using "Welch Allyn" (oral/rectal), Covidien (tympanic) and ARC InstaTempMD (non-touch, infrared) in degrees Celcius and will be compared with three consecutive measurements with each thermometer. | Participant will only be required to attend one visit which will last up to a maximum of 30 minutes for the duration of the study.
  Compare the compendia thermometers in each age range to the InstaTemp MD to determine average clinical bias.

SECONDARY OUTCOMES:
Mean Comparison Analysis. Temperature measurements using "Welch Allyn" (oral/recta.), Covidien (tympanic) and ARC InstaTemp MD (non-touch, infrared) in degrees Celcius and will be compared with three consecutive measurements with each thermometer. | Participant will only be required to attend one visit which will last up to a maximum of 30 minutes for the duration of the study.
  To determine the precision of the InstaTemp MD compared to the compendia thermometers based on three consecutive measurements with each thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: Judy van Stralen, MD FRCPC, Principal Investigator — Center for Pediatric Excellence
Locations (2):
- Canada (2):
  - Center for Pediatric Excellence, Ottawa, Ontario
  - Agoo Children's Health and Wellness Centre, Laval, Quebec

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03147534/Prot_000.pdf